CLINICAL TRIAL: NCT01193933
Title: Multicenter Clinical Trial for Adult Ph-negative ALL. Evaluation of the Impact of the Prolonged L-asparaginase Therapy During Continuous Treatment With Modification of Cytostatic Drugs Doses Depending on Myelosuppression Severity.
Brief Title: Multicenter Clinical Trial for Adult Ph-negative ALL. Non-intensive But Non-iterruptive Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, MD PhD, National Research Center for Hematology, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL-2009
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Ph-negative Adult Acute Lymphoblastic Leukemia
Keywords: adult ALL; Ph-negative; dexamethasone; L-asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: autologous HSCT — T-cell ALL patients recieve late consolidation with BEAM conditioning and stem cell support

SUMMARY:
1. evaluation of blast clearance in b/m after 7 days of prednisolone prephase and the efficacy of its substitution by dexamethasone if blast count is 25% and more
2. feasibility for adults of "no interruptions" protocol with 8 weeks induction and 14 weeks consolidation followed by 2-years maintenance.
3. tolerability and efficacy in adults of the prolonged L-asparaginase application (total proposed dose 560.000 IU)
4. feasibility and efficacy of autologous stem cell transplantation for T-cell ALL

DETAILED DESCRIPTION:
1. The blast count in b/m after 7 days of prednisolone >25% was shown in 64% of patients. The substitution of prednisolone by dexamethasone did not influence survival.
2. "no interruptions" induction was performed in 48% of patients.
3. In 19% of patients the L-asparaginase therapy was stopped due to toxicity.
4. Autologous stem cell transplantation was done in 20% of T-cell ALL patients.

ELIGIBILITY:
Inclusion Criteria:

* Ph-negative precursors ALL
* age 15-55 years
* nontreated
* Eastern Cooperative Oncology Group criterion status 0-3

Exclusion Criteria:

* B-mature ALL
* Ph-positivity
* pretreatment
* Eastern Cooperative Oncology Group criterion status 4

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 321 (Estimated)
Dates: Start 2008-11; Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of adult ALL patients who tolerated the non-interrupted treatment | 3 years
  Number of patients who finished the protocol without any deviation, who were off the protocol due to toxicity, in whom the treatment schedule was modified and respectively the antileukemia efficacy in those subgroups

SECONDARY OUTCOMES:
Toxicity of prolonged L-asparaginase in adult patients | 3 years
  Number of patients who tolerated the scheduled L-asparaginase by dose and time sequence, proportion of patients shifted to PEG-asparaginase, in whom L-asparaginase was stopped and, respectively, the survival without leukemia of those patients

CONTACTS AND LOCATIONS:
Overall Officials: Valeri G Savchenko, Professor, Study Chair — National Research Center for Hematology
Locations (1):
- Russian Acute Lymphoblastic Leukemia Study group, Moscow, Russia

REFERENCES:
- [Derived] Parovichnikova EN, Troitskaya VV, Gavrilina OA, Sokolov AN, Kokhno AV, Klyasova GA, Kuzmina LA, Galstyan GM, Makhinya SA, Latyshkevich OA, Kaporskaya TS, Lapin VA, Chabaeva YA, Kulikov SM, Savchenko VG; for Russian Acute Lymphoblastic Leukemia group. The outcome of Ph-negative acute lymphoblastic leukemia presenting during pregnancy and treated on the Russian prospective multicenter trial RALL-2009. Leuk Res. 2021 May;104:106536. doi: 10.1016/j.leukres.2021.106536. Epub 2021 Feb 14. PMID 33676165
- [Derived] Parovichnikova E, Troitskaya V, Sokolov A, Gavrilina O, Akhmerzaeva Z, Kuzmina L, Kliasova G, Chabaeva J, Kulikov S, Bondarenko S, Baranova O, Samoilova O, Kaplanov K, Minaeva N, Savchenko V; Russian Acute Lymphoblastic Leukemia Group. Can Less Intensive Chemotherapy and an Autotransplant Cure Adult T-Cell Acute Lymphoblastic Leukemia? Acta Haematol. 2020;143(2):131-139. doi: 10.1159/000502435. Epub 2019 Oct 9. PMID 31597157
- [Derived] Piskunova IS, Obukhova TN, Parovichnikova EN, Kulikov SM, Troitskaya VV, Gavrilina OA, Savchenko VG. Structure and significance of cytogenetic abnormalities in adult patients with Ph-negative acute lymphoblastic leukemia. Ter Arkh. 2018 Aug 17;90(7):30-37. doi: 10.26442/terarkh201890730-37. PMID 30701920
- [Derived] Parovichnikova EN, Troitskaya VV, Sokolov AN, Bondarenko SN, Gavrilina OA, Baskhaeva GA, Biderman BV, Lukyanova IA, Kuz'mina LA, Klyasova GA, Kravchenko SK, Gribanova EO, Zvonkov EE, Akhmerzaeva ZK, Baranova OY, Kaporskaya TS, Ryltsova TV, Zotina EN, Zinina EE, Samoilova OS, Kaplanov KD, Gavrilova LV, Konstantinova TS, Lapin VA, Pristupa AS, Eluferyeva AS, Obukhova TN, Piskunova IS, Gal'tseva IV, Dvirnyk VN, Rusinov MA, Kulikov SM, Savchenko VG. [Adult B-cell acute lymphoblastic leukemias: Conclusions of the Russian prospective multicenter study ALL-2009]. Ter Arkh. 2017;89(7):10-17. doi: 10.17116/terarkh201789710-17. Russian. PMID 28766535
- [Derived] Parovichnikova EN, Kuzmina LA, Mendeleeva LP, Klyasova GA, Troitskaya VV, Sokolov AN, Akhmerzaeva ZK, Kravchenko SK, Gribanova EO, Zvonkov EE, Bondarenko SN, Baranova OY, Ryltsova TV, Gavrilova LV, Zinina EE, Pristupa AS, Kaporskaya TS, Minaeva NV, Samoilova OS, Konstantinova TS, Lapin VA, Kaplanov KD, Kryuchkova IV, Nizamutdinova AS, Klimovich AV, Borisenkova EA, Moskov VI, Gaponova TV, Obukhova TV, Galtseva IV, Rusinov MA, Kulikov SM, Savchenko VG. [Autologous hematopoietic stem cell transplantation as late high-dose consolidation in adult patients with T-cell lymphoblastic leukemias: Results of a Russian multicenter study]. Ter Arkh. 2015;87(7):15-25. doi: 10.17116/terarkh201587715-25. Russian. PMID 26390721